CLINICAL TRIAL: NCT06694350
Title: Safety and Efficacy of Pembrolizumab in Combination with Flutamide Treatment for Advanced/Recurrence / Metastasis Head and Neck Squamous Cell Carcinoma: a Single-arm Clinical Study Trial
Brief Title: Pembrolizumab in Combination with Flutamide Treatment for Recurrence / Metastasis HNSCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KF20240822
Record Dates: First submitted 2024-10-31; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab+Flutamide (Experimental): Pembrolizumab 200mg ivgtt once +Flutamide 250mg，Q8h
  Interventions: Drug: Pembrolizumab+Flutamide

INTERVENTIONS:
Drug: Pembrolizumab+Flutamide — Pembrolizumab 200mg ivgtt once +Flutamide 250mg，Q8h

SUMMARY:
This study is a single center, single arm clinical trial for newly diagnosed patients with locally advanced head and neck squamous cell carcinoma. The main purpose is to evaluate the efficacy and safety of flutamide combined with standard immunotherapy for advanced / recurrent head and neck squamous cell carcinoma.

In our previous study, we found that AR can affect the occurrence and development of tumors by regulating the differentiation of cd8+t cells. We used three different castration drugs (flutamide, goserelin and abiraterone) in animal models to treat primary and tumor bearing head and neck squamous cell carcinoma mice respectively, and found that castration treatment could significantly inhibit the tumor growth of head and neck squamous cell carcinoma. In addition, in animal models, we compared the efficacy of the combination of castration therapy and low-dose cisplatin with that of the existing first-line chemotherapy drug cisplatin, and found that the combination of castration therapy and low-dose cisplatin can significantly improve the treatment effect of head and neck squamous cell carcinoma and reduce the adverse reactions brought by the drug. Therefore, we infer that flutamide combined with standard immunotherapy can fully inhibit the growth of HNSCC and improve the prognosis of HNSCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, ≤ 85 years old
2. Histologically or cytologically proven squamous cell carcinoma of the head and neck; Patients diagnosed with head and neck squamous cell carcinoma with stage III and IV A without distant metastasis according to AJCC staging (8th editon), including squamous cell carcinoma of oropharyngeal (P16-), oral cavity, hypopharyngeal and larynx
3. Measurable primary lesions per RECIST 1.1 criteria
4. Treatment-naive patients without any previous disease-related therapy (except for diagnostic biopsies on primary lesions)
5. ECOG performance status of 0 or 1
6. Unresectable primary, recurrent, and / or metastatic HNSCC
7. No active autoimmune disease
8. No concurrent malignancy
9. Life expectancy is estimated to be over 3 months
10. Have sufficient tumour tissue samples available for CPS PD-L1 immunohistochemical examination (22C3 DAKO)
11. No abvious signs of hematological disorders, ANC≥1.5×109 /L, platelets ≥100×109 /L, Hb≥ 90 g/L,WBC ≥3.0×109 /L before enrollment, no blood transfusion and bleeding tendency within 7 days
12. ALT,AST and ALP ≤ 2.5 × upper limit of normal (ULN); Serum bilirubin ≤ 1.5 × ULN, for patients with known Gilbert disease, serum bilirubin ≤ 3 x ULN
13. Serum creatinine ≤1.5 or creatinine clearance>50 mL/min
14. HPV status determined by p16 IHC, in situ hybridization, or by polymerase chain reaction-based assays
15. Able to understand this study, patient and (or) legal representative voluntarily agree to participate in this trial and sign informed consent

Exclusion Criteria:

1. Patients who are suitable for local treatment and have the intention of local treatment
2. Received systemic treatment with Chinese patent drugs with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin) within 2 weeks before the first administration
3. Patients with tumor progression after previous treatment with flutamide analogues (antiandrogens)
4. Other malignant tumors occurred within 5 years or suffered from at the same time in the current period, except for cured non melanoma skin cancer or other tumors / cancers that have undergone radical treatment and have no signs of disease for at least 5 years;
5. According to the criteria of common adverse event terminology (NCI ctcaev5.0), there was peripheral neuropathy ≥ grade 2
6. With known active central nervous system metastasis (CNS) and / or cancerous meningitis
7. Subjects who did not recover from any acute effects of previous surgery, chemotherapy or radiotherapy, i.e. did not fall to grade ≤ 1 (NCI ctcaev5.0) (excluding hair loss). Chronic late toxicity from previous radiotherapy and / or surgery is allowed if nutritional status is stable
8. Any component of the study drug or preparation has led to severe allergic reactions, including known severe allergic reactions to flutamide and (NCI ctcaev5.0 ≥ grade 3)
9. Have received anti-tumor drug treatment (such as chemotherapy, hormone therapy, immunotherapy, antibody therapy, radiotherapy, etc.) within 4 weeks or 4 weeks before the first administration, except for palliative radiotherapy for bone to reduce pain
10. Major surgery within 4 weeks before the first dose or expected during this study
11. Immunosuppressive drugs were required 2 weeks or within 2 weeks before the first dose or during the study
12. Subjects who are known to have active, or have a history of autoimmune disease that may recur
13. Subjects with known history of interstitial lung disease, non infectious pneumonia, or high suspicion of interstitial lung disease
14. Hepatitis B or C virological examination meets any of the following requirements at the time of screening:

    1. HBsAg is positive, and the titer of hepatitis B virus deoxyribonucleic acid (HBV DNA) in peripheral blood is ≥ 104 copies /ml or ≥ 2000 iu/ml;
    2. HCV antibody was positive, and HCV-RNA was higher than the detection limit of the analytical method;
15. Within 2 weeks or 2 weeks before the first administration, the subject had active infection or uncontrollable infection requiring systemic treatment (except simple urinary tract infection or upper respiratory tract infection)
16. Serous cavity effusion with clinical symptoms requiring clinical intervention or stabilization time less than 4 weeks
17. Diabetes mellitus (fasting blood glucose ≥ 10mmol/l) or hypertension (systolic blood pressure ≥ 160mmhg and / or diastolic blood pressure ≥ 100mmhg) with severe medical diseases, such as grade III or above cardiac dysfunction (New York Heart Association [nyha]), ischemic heart disease (such as myocardial infarction or angina pectoris) and other cardiovascular diseases, or a history of myocardial infarction within 3 months before the first administration, and still poorly controlled after drug treatment (fasting blood glucose ≥ 10mmol/l) or poorly controlled hypertension (systolic blood pressure ≥ 160mmhg and / or diastolic blood pressure ≥ 100mmhg)
18. Medical or psychiatric history or history of laboratory abnormalities that may interfere with the interpretation of the results
19. Subjects are currently enrolled in the study of other investigational devices or investigational drugs, or are less than or equal to 4 weeks away from the discontinuation of other investigational drugs or investigational devices
20. Subjects were known to have alcohol or drug addiction
21. Subjects have other conditions that may affect their compliance with the protocol and evaluation of research indicators, and are not suitable to participate in the study

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 4 years
  The Progression-Free-Survival of Interventions group

SECONDARY OUTCOMES:
ORR | Up to 4 years
  The Objective Response Rate of Intervention group
DOR | Up to 4 years
  The Disease Control Rate of intervention group
OS | Up to 4 years
  The overall survival of paticipated patients